CLINICAL TRIAL: NCT02886936
Title: Immediate Fit Using Innovative Technology Transtibial & Transfemoral Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: iFIT Prosthetics, LLC (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 815654; 2R42AG050430 (NIH); 2SB1AG050430-06 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Amputation
Keywords: transtibial; transfemoral

STUDY DESIGN:
Intervention Model Description: single-group pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transtibial Testing (Experimental): This is a feasibility and effectiveness study to assess the iFIT transtibial prosthesis as a viable alternative to a traditional prosthesis. We also hope to gain information that will influence future design iterations.
  Interventions: Device: iFIT Transtibial Prosthesis
- Transfemoral Testing (Experimental): This is a feasibility and effectiveness study to assess the iFIT transfemoral prosthesis as a viable alternative to a traditional prosthesis. We also hope to gain information that will influence future design iterations.
  Interventions: Device: iFIT Transfemoral Prosthesis

INTERVENTIONS:
Device: iFIT Transtibial Prosthesis — Transtibial amputee volunteers will be fit with the iFIT device and instructed on its use. Patient will wear the iFIT device for a two week time period according to a provided wear schedule. At the end of this time patient will rate it for comfort, stability and ease of use.
  Arms: Transtibial Testing
Device: iFIT Transfemoral Prosthesis — Transfemoral amputee volunteers will be fit with the iFIT device and instructed on its use. Patient will wear the iFIT device for a two week time period according to a provided wear schedule. At the end of this time patient will rate it for comfort, stability and ease of use.
  Arms: Transfemoral Testing

SUMMARY:
iFIT Prosthetics, LLC® created and commercialized a modular, immediate fit, fully adjustable, prosthetic system suitable for mass production using high strength injection molded polymer materials. The aim of this project is to assess the design, user satisfaction and feasibility of this device. The investigators will be fitting transtibial and transfemoral amputees with the iFIT prosthetic system. Patients will wear the device for 2 weeks in order to compare the device to their own prosthetic (if they currently have one). They will report any device breakages or adverse events. They will also fill out a questionnaire to determine if the iFIT prosthetic is a feasible option for treating patients with limb loss.

ELIGIBILITY:
Inclusion Criteria:

* transtibial or transfemoral level of amputation
* functional ambulator with or without a cane
* six months or more since amputation.

Exclusion Criteria:

* patient have skin ulcerations on the residual limb
* have other central nervous system disorders such as strokes and brain injuries that interfere with safe ambulation and gait testing
* severe phantom or limb pain
* weight over 260 lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dillingham, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Dillingham T, Kenia J, Shofer F, Marschalek J. A Prospective Assessment of an Adjustable, Immediate Fit, Transtibial Prosthesis. PM R. 2019 Nov;11(11):1210-1217. doi: 10.1002/pmrj.12133. Epub 2019 Apr 1. PMID 30734517
- [Result] McCloskey C, Kenia J, Shofer F, Marschalek J, Dillingham T. Improved Self-Reported Comfort, Stability, and Limb Temperature Regulation with an Immediate Fit, Adjustable Transtibial Prosthesis. Arch Rehabil Res Clin Transl. 2020 Dec;2(4):100090. doi: 10.1016/j.arrct.2020.100090. Epub 2020 Nov 2. PMID 33381750
- [Result] Dillingham TR, Kenia JL, Shofer FS, Marschalek JS. A Prospective Assessment of an Adjustable, Immediate Fit, Subischial Transfemoral Prosthesis. Arch Rehabil Res Clin Transl. 2022 May 2;4(3):100200. doi: 10.1016/j.arrct.2022.100200. eCollection 2022 Sep. PMID 36123976

RESULTS

PARTICIPANT FLOW:
Groups:
- Transtibial Testing Study 1: This is a feasibility and effectiveness study to assess the iFIT transtibial prosthesis as a viable alternative to a traditional prosthesis. We also hope to gain information that will influence future design iterations.
  iFIT Transtibial Prosthesis: Transtibial amputee volunteers will be fit with the iFIT device and instructed on its use. Patient will wear the iFIT device for a two week time period according to a provided wear schedule. At the end of this time patient will rate it for comfort, stability and ease of use.
- Transtibial Testing Study 2 (Follow Up): This is a follow up feasibility and effectiveness study to assess the iFIT transtibial prosthesis as a viable alternative to a traditional prosthesis. We also hope to gain information that will influence future design iterations.
  iFIT Transtibial Prosthesis: Transtibial amputee volunteers will be fit with the iFIT device and instructed on its use. Patient will wear the iFIT device for a two week time period according to a provided wear schedule. At the end of this time patient will rate it for comfort, stability and ease of use.
Period: Overall Study
Arm/Group | Transtibial Testing Study 1 | Transtibial Testing Study 2 (Follow Up) | Transfemoral Testing
Started | 26 (This is from our first and follow up study on the transtibial.) | 27 | 18
Completed | 22 | 24 | 18
Not Completed | 4 | 3 | 0
Not completed — Lost to Follow-up | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Transtibial and Transfemoral subjects that enrolled in the study.
Groups:
- Transtibial Testing Study 2: This is a follow up feasibility and effectiveness study to assess the iFIT transtibial prosthesis as a viable alternative to a traditional prosthesis. We also hope to gain information that will influence future design iterations.
  iFIT Transtibial Prosthesis: Transtibial amputee volunteers will be fit with the iFIT device and instructed on its use. Patient will wear the iFIT device for a two week time period according to a provided wear schedule. At the end of this time patient will rate it for comfort, stability and ease of use.
- Total: Total of all reporting groups
Arm/Group | Transtibial Testing Study 1 | Transtibial Testing Study 2 | Transfemoral Testing | Total
Number analyzed (Participants) | 26 | 27 | 18 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 12 | 55
  >=65 years | 4 | 6 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10.2) | 55 (13.2) | 59.4 (7) | 54.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 2 | 11
  Male | 22 | 22 | 16 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/ not Hispanic | 12 | 11 | 10 | 33
  Race/Ethnicity: Hispanic/ Latino | 0 | 3 | 2 | 5
  Race/Ethnicity: African American/Black | 14 | 13 | 6 | 33
  Race/Ethnicity: Asian/ Pacific Islander | 0 | 0 | 0 | 0
  Race/Ethnicity: Other | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 27 | 18 | 71

OUTCOME MEASURES:

1. Primary Outcome: Prosthetic Comfort and Utility Questionnaire (Version 1)
Description: This questionnaire is based off of the Prosthetic Evaluation Questionnaire; it involves questions taken from the original that focus on comfort, satisfaction and utility of a prosthetic socket. We used numeric values from 1 (Poor) through 5 (Excellent) for evaluation.
  This version featured seven questions for a total of 35 points possible and the lowest score being 7 (higher scores are better). Scores are reported as total with standard deviations.
Time Frame: 2 weeks
Population: Persons completing the two week trial from the first cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 22
score on a scale
  Conventional Prosthesis | 25.52 (6.8)
  iFIT Prosthesis | 29.33 (4.51)

2. Primary Outcome: Prosthetic Comfort and Utility Questionnaire (Version 2)
Description: This questionnaire is based off of the Prosthetic Evaluation Questionnaire; it involves questions taken from the original that focus on comfort, satisfaction and utility of a prosthetic socket. We used numeric values from 1 (Poor) through 5 (Excellent) for evaluation.
  This version features fourteen questions for a total of 70 points total, with the lowest score being 14. Higher scores are better. Scores are reported as total with standard deviations.
Time Frame: 2 weeks
Population: Transtibial participants that returned for 2 week follow up in the second cohort of subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transtibial Testing Study 2 (Follow Up)
Number analyzed (Participants) | 24
score on a scale
  iFIT Prosthesis | 29 (4.5)
  Conventional Prosthesis | 25.4 (6.8)

3. Primary Outcome: Prosthetic Comfort and Utility Evaluation (Version 3)
Description: This questionnaire is based off of the Prosthetic Evaluation Questionnaire; it involves questions taken from the original that focus on comfort, satisfaction and utility of a prosthetic socket. We used numeric values from 1 (Poor) through 5 (Excellent) for evaluation.
  This version features ten questions for a total of 50 points possible, with the lowest score being 10. Higher scores are better. Scores are reported as total with standard deviations.
Time Frame: 2 weeks
Population: Participants with transfemoral limb loss that completed the two week follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transfemoral Testing
Number analyzed (Participants) | 18
score on a scale
  iFIT Prosthesis | 40.9 (7.2)
  Conventional Prosthesis | 32.8 (10.2)

4. Secondary Outcome: Number of Participants With Device Related Adverse Events
Description: We will record any unfavorable events such that occur including: skin irritation, skin breakdown, falls, or mechanical failures.
Time Frame: 2 weeks
Population: Participant completing the study
Measure: Count of Participants; unit: Participants
Arm/Group | Transtibial Testing Study 1 | Transtibial Testing Study 2 (Follow Up) | Transfemoral Testing
Number analyzed (Participants) | 22 | 24 | 18
Participants
  Serious adverse event: Fall, device breakage, limb ischemia | 0 | 0 | 0
  Minor adverse event: skin irritation or minor skin breakdown | 2 | 0 | 0
  NO Adverse Events | 20 | 24 | 18

5. Secondary Outcome: Gait Analysis- Walking Speed
Description: Gait speed is the time one takes to walk a specified distance on level surfaces over a short distance.
Time Frame: two weeks
Population: Persons from the first cohort (transtibial testing study 1) that completed the two week trial and had unilateral amputation. Cohort two was not tested. Persons with transfemoral amputation were not tested due to a difference in knees between testing conditions.
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 17
m/s
  Walking Speed Prosthetic Side - iFIT | .98 [.98 to 1]
  Walking Speed Prosthetic Side - Conventional | .98 [.97 to 1]
  Walking Speed Sound Side- iFIT | .98 [.97 to 1]
  Walking Speed Sound Side - Conventional | .98 [.97 to 1]

6. Secondary Outcome: Internal Socket Pressure
Description: Fujifilm prescale was placed on five specific places on the outside of the participant's liner. They then ambulated for two minutes. The paper was removed and average pressure was recorded. This was completed for both sockets.
Time Frame: Two weeks
Population: This was completed on the first cohort for transtibial testing study 1. Testing was not completed on the second cohort or the transfemoral cohort.
Measure: Mean (Standard Deviation); unit: p/si
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 22
p/si
  iFIT Overall Avg Pressure | 17.3 (2.3)
  Conventional Overall Avg Pressure | 19.3 (3.7)
  iFIT Tibial Avg Pressure | 18 (4.2)
  Conventional Tibial Avg Pressure | 22 (3.7)
  iFIT Medial Avg Pressure | 15.5 (2.6)
  Conventional Medial Avg Pressure | 16.3 (5.5)
  iFIT Posterior Avg Pressure | 16.5 (3.6)
  Conventional Posterior Avg Pressure | 18.1 (7.5)
  iFIT Bottom Avg Pressure | 20 (3.5)
  Conventional Bottom Avg Pressure | 20.5 (4.1)
  iFIT Lateral Avg Pressure | 16.5 (4.8)
  Conventional Lateral Avg Pressure | 19.3 (4.9)

7. Secondary Outcome: Gait Analysis - Double Support
Description: Double support is the amount of time that both feet are touching the ground during walking. A faster gait will correlate with lower values since less time is spent with both feet on the ground; consequently, a slower gait will yield higher values.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 17
seconds
  Double Support Prosthetic Side- iFIT | .37 [.36 to .38]
  Double Support Prosthetic Side - Conventional | .36 [.34 to .36]
  Double Support Sound Side- iFIT | .37 [.37 to .38]
  Double Support Sound Side- Conventional | .35 [.34 to .36]

8. Secondary Outcome: Gait Analysis - Limp Index
Description: Limp index is a temporal parameter used in gait analysis to describe symmetry when walking. For a symmetric walk, the limp index is exactly one; values significantly higher or lower than 1 denote greater asymmetry. It is calculated by using the total support (single + double) for the current foot divided by the total support for the opposite foot.
Time Frame: 2 weeks
Population: Participants from the first cohort (transtibial testing study 1) that completed the two week trial and had unilateral amputation. Persons in cohort two were not tested. Persons for the transfemoral testing were not tested as the componentry (prosthetic knees) were markedly different.
Measure: Mean (95% Confidence Interval); unit: Index
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 17
Index
  Limp Index Prosthetic Side - iFIT | .99 [.96 to 1]
  Limp Index Prosthetic Side- Conventional | .97 [.95 to 1]
  Limp Index Sound Side- iFIT | 1.01 [1 to 1.04]
  Limp Index Sound Side - Conventional | 1.03 [1.01 to 1.05]

9. Secondary Outcome: Gait Analysis - Stride Length
Description: Stride length is the distance between successive points of initial contact of the same foot. Right and left stride lengths are normally equal.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 17
meters
  Stride Length Prosthetic Side - iFIT | 1.22 [1.21 to 1.25]
  Stride Length Prosthetic Side - Conventional | 1.22 [1.21 to 1.24]
  Stride Length Sound Side - iFIT | 1.22 [1.21 to 1.25]
  Stride Length Sounds Side - Conventional | 1.21 [1.20 to 1.24]

10. Secondary Outcome: Gait Analysis Stance Phase
Description: Begins when the foot first touches the ground and ends when the same foot leaves the ground. Expressed as a percentage of the total gait cycle.
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of gait cycle
Arm/Group | Transtibial Testing Study 1
Number analyzed (Participants) | 17
Percentage of gait cycle
  Stance Phase- Prosthetic Side iFIT Avg | 64.3 [63.3 to 64.6]
  Stance Phase- Prosthetic Side Conventional Avg | 63.4 [62.4 to 63.7]
  Stance Phase- Sound Side iFIT Avg | 65.2 [64.6 to 65.9]
  Stance Phase - Sound Side Conventional Avg | 65 [64.3 to 65.6]

11. Secondary Outcome: Residual Limb Circumference Measurements to Internal Socket Diameter
Description: The subject's residual limb was measured at the proximal 1/3, midpoint and distal 1/3 while wearing their liner and on skin. This was compared to their internal socket circumference.
Time Frame: Same Day
Population: Only the transfemoral subjects were analyzed. This outcome measure was added after the transtibial subjects were tested.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Transfemoral Testing
Number analyzed (Participants) | 18
cm
  Avg Circumference No Liner Proximal 1/3 | 51.7 (7.2)
  Avg Circumference No Liner Mid Point | 47.2 (7.7)
  Avg Circumference No Liner Distal 1/3 | 40.6 (7)
  Avg Circumference WITH Liner Proximal 1/3 | 53.6 (7.2)
  Avg Circumference WITH Liner Mid Point | 47.7 (6.1)
  Avg Circumference WITH Liner Distal 1/3 | 41.3 (5.9)
  Avg Internal Socket Circumference Proximal 1/3 | 46.3 (5.3)
  Avg Internal Socket Circumference Mid Point | 40.5 (4.9)
  Avg Internal Socket Circumference Distal 1/3 | 35.7 (5.6)
  Avg Difference Between Limb and Socket While Wearing Liner Proximal 1/3 | 7.3 (3.6)
  Avg Difference Between Limb and Socket While Wearing Liner Mid Point | 7.2 (3.9)
  Avg Difference Between Limb and Socket While Wearing Liner Distal 1/3 | 5.6 (4.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Serious events were recorded during the follow up. They were obtained by visual inspection of the skin and prosthesis, and through verbal report from the participant.
Groups:
- Transtibial Testing 2(Follow Up): This is a follow up feasibility and effectiveness study to assess the iFIT transtibial prosthesis as a viable alternative to a traditional prosthesis. We also hope to gain information that will influence future design iterations.
  iFIT Transtibial Prosthesis: Transtibial amputee volunteers will be fit with the iFIT device and instructed on its use. Patient will wear the iFIT device for a two week time period according to a provided wear schedule. At the end of this time patient will rate it for comfort, stability and ease of use.
Arm/Group | Transtibial Testing | Transtibial Testing 2(Follow Up) | Transfemoral Testing
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/18
Other Adverse Events (participants affected / at risk) | 2/26 | 0/27 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transtibial Testing (N=26) | Transtibial Testing 2(Follow Up) (N=27) | Transfemoral Testing (N=18)
Skin Breakdown (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Skin breakdown

LIMITATIONS AND CAVEATS:
Participants that entered the study may have been dissatisfied with their current prosthesis.

This research was conducted at a single location.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT02886936/Prot_SAP_000.pdf